CLINICAL TRIAL: NCT04172623
Title: Evaluating the Feasibility and Efficacy of a Real-time Smoking Intervention Using Wearable Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Patterson Trust Mentored Research Award: Clinical, Health Services and Policy Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000024740
Record Dates: First submitted 2019-07-08; First posted 2019-11-21 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: Parallel group randomized trial design comparing smoking outcomes when receiving standard treatment vs. standard treatment plus real-time smoking intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-Time Smoking Intervention (Experimental): Adult smokers will use wearable technology in order to receive real-time feedback as a smoking intervention in addition to standard treatment.
  Interventions: Behavioral: Real-Time Smoking Intervention; Behavioral: Standard Treatment
- Standard Treatment (Active Comparator): Adult smokers will receive standard outpatient tobacco treatment.
  Interventions: Behavioral: Standard Treatment

INTERVENTIONS:
Behavioral: Real-Time Smoking Intervention — Adult smokers will use wearable technology in order to receive real-time feedback as a smoking intervention in addition to standard treatment.
  Arms: Real-Time Smoking Intervention
Behavioral: Standard Treatment — Adult smokers will receive standard outpatient tobacco treatment.

SUMMARY:
This study will use wearable technology to test the feasibility and efficacy of delivering a novel real-time smoking intervention to improve standard tobacco treatment.

DETAILED DESCRIPTION:
The goals of this project include evaluating the feasibility, acceptability, and helpfulness of the real-time smoking intervention and to assess the preliminary efficacy of the real-time intervention as an adjunct to standard tobacco treatment. Rates of adherence, participant satisfaction, and perceived usefulness will be evaluated through post-treatment interviews and ratings. Biochemically confirmed 7-day point prevalence abstinence will be compared between the experimental and control groups at the end of treatment (week 8).

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Able to read English
* Cigarette smoker
* Seeking smoking cessation treatment

Exclusion Criteria:

* Serious psychiatric or medical condition
* Unable or unwilling to complete study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krysten Bold, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real-Time Smoking Intervention | Standard Treatment
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real-Time Smoking Intervention | Standard Treatment | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (10.3) | 57.9 (9.4) | 56.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Self-report data on sex was missing for N=4 participants, N=2 in each condition.
  Participants
    number analyzed (Participants) | 27 | 27 | 54
    Female | 17 | 14 | 31
    Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Self-reported ethnicity data were missing for N=4 participants, N=2 in each condition.
  Participants
    Hispanic or Latino | 3 | 5 | 8
    Not Hispanic or Latino | 24 | 22 | 46
    Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 14 | 17 | 31
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in Cigarettes
Description: Self-reported cigarette use (Timeline follow-back data) during the 8-week study to estimate effect sizes between groups.
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Real-Time Smoking Intervention | Standard Treatment
Number analyzed (Participants) | 29 | 29
cigarettes per day | 10.2 (12.2) | 7.7 (6.5)

2. Secondary Outcome: % Days Abstinent From Cigarettes
Description: Timeline follow-back data will be collected to determine the % of days abstinent from cigarettes.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Real-Time Smoking Intervention | Standard Treatment
Number analyzed (Participants) | 29 | 29
percentage of days | 12.4 (27.2) | 6.9 (14.6)

ADVERSE EVENTS:
Time Frame: 8 week treatment period
Arm/Group | Real-Time Smoking Intervention | Standard Treatment
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT04172623/Prot_SAP_000.pdf